CLINICAL TRIAL: NCT04763811
Title: Acceptability Study of Sensor in Elderly People's House Living Alone
Brief Title: Acceptability Study of Sensor in Elderly People's House Living Alone (Fragility Box)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Saint Etienne School of Mine (Other); Eovi Mcd Mutuelle (Unknown); Gerontopole Auvergne Rhone-Alpes (AURA) (Other)
Responsible Party: Sponsor
Other Study IDs: GA-2021-01
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Aging
Keywords: sensors; acceptability; qualitative study; autonomous; elderly people; prevention; Autonomy loss
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older 65 people: Older 65 people who live alone in their house will be included. They will have focus groups and Individual interviews.
  Interventions: Other: Focus groups; Other: Individual interviews

INTERVENTIONS:
Other: Focus groups — discussion between participants about representations of health, dependance, fragility, and new technologies
Other: Individual interviews — Discussion between the searcher and the participant about representations of captors, discretion of captors, wish about feed-backs of captors

SUMMARY:
The Fragility box is a project lead by Mines de Saint-Etienne, Gérontopôle Auvergne-Rhône-Alpes (AURA) and Eovi Mcd Mutually to prevent autonomy loss in the elderly dwelling population. With non-intrusive sensors installed in their residence, it is possible to monitor and forecast the frail state of elderly people living alone. The current study focuses on the technical feasibility of the project and the acceptability of these types of devices within the elderly's home. About ten participants have volunteered to be a part of this study. Therefore, they had the sensors installed at their home for a 12 months duration. A qualitative study with focus groups and individual interviews are carried out to evaluate the project: user satisfaction, expectations, and fears.

DETAILED DESCRIPTION:
This research tend to study the acceptability of captors which can measure the evolution of autonomy of older 65 people.

ELIGIBILITY:
Inclusion Criteria:

* People living alone
* Autonomous person

Exclusion Criteria:

* Person with a neurological disease
* Person under guardianship or curatorship

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older 65 people who live alone in their own house
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Analysis representations of health/fragility and new technologies | Months:6
  Measured by focus groups results.

SECONDARY OUTCOMES:
Analysis Representations of health and frailties ; and new technologies Acceptability of sensors | Months:6
  Measured by individual interviews results.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Augusto, Study Director — augusto@emse.fr
Locations (1):
- Gérontopole AURA, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No